CLINICAL TRIAL: NCT05367440
Title: A Multi-arm, Open-label Phase I/IIa Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of AZD5305 in Combination With New Hormonal Agents in Patients With Metastatic Prostate Cancer (PETRANHA)
Brief Title: Study of AZD5305 When Given in Combination With New Hormonal Agents in Patients With Metastatic Prostate Cancer
Acronym: PETRANHA
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9720C00003; 2023-508536-64-00 (Registry Identifier: CTIS); 2021-006289-19 (EudraCT Number)
Record Dates: First submitted 2022-04-19; First posted 2022-05-10 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Prostate Cancer
Keywords: PETRANHA; AZD5305; New Hormonal Agents
MeSH Terms: conditions — Prostatic Neoplasms | interventions — AZD5305; enzalutamide; Abiraterone Acetate; darolutamide; apalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1 (AZD5305 in combination with enzalutamide) (Experimental): Patients will receive an oral dose of AZD5305 and Enzalutamide once daily until disease progression, initiation of alternative anticancer therapy, unacceptable toxicity, withdrawal of consent, or other reasons to discontinue study treatment occur.
  Interventions: Drug: AZD5305; Drug: Enzalutamide
- Arm 2 (AZD5305 in combination with abiraterone acetate) (Experimental): Patients will receive an oral dose of AZD5305 and Abiraterone Acetate once daily until disease progression, initiation of alternative anticancer therapy, unacceptable toxicity, withdrawal of consent, or other reasons to discontinue study treatment occur.
  Interventions: Drug: AZD5305; Drug: Abiraterone Acetate
- Arm 3 (AZD5305 in combination with darolutamide) (Experimental): Patients will receive an oral dose of AZD5305 once daily and Darolutamide twice daily until disease progression, initiation of alternative anticancer therapy, unacceptable toxicity, withdrawal of consent, or other reasons to discontinue study treatment occur.
  Interventions: Drug: AZD5305; Drug: Darolutamide
- Arm 4 (AZD5305 in combination with apalutamide) (Experimental): Patients will receive an oral dose of AZD5305 and Apalutamide once daily until disease progression, initiation of alternative anticancer therapy, unacceptable toxicity, withdrawal of consent, or other reasons to discontinue study treatment occur.
  Interventions: Drug: Apalutamide

INTERVENTIONS:
Drug: AZD5305 — Patients will receive an oral dose of AZD5305 once daily
  Arms: Arm 1 (AZD5305 in combination with enzalutamide); Arm 2 (AZD5305 in combination with abiraterone acetate); Arm 3 (AZD5305 in combination with darolutamide)
Drug: Enzalutamide — Patients will receive an oral dose of Enzalutamide once daily
  Other Names: Xtandi
  Arms: Arm 1 (AZD5305 in combination with enzalutamide)
Drug: Abiraterone Acetate — Patients will receive an oral dose of Abiraterone Acetate once daily
  Other Names: Zytiga
  Arms: Arm 2 (AZD5305 in combination with abiraterone acetate)
Drug: Darolutamide — Patients will receive an oral dose of Darolutamide twice daily
  Other Names: Nubeqa
  Arms: Arm 3 (AZD5305 in combination with darolutamide)
Drug: Apalutamide — Patients will receive an oral dose of Apalutamide once daily
  Other Names: Erleada
  Arms: Arm 4 (AZD5305 in combination with apalutamide)

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and preliminary efficacy of AZD5305 when given in combination with new hormonal agents (NHAs) in patients with Metastatic Prostate Cancer.

DETAILED DESCRIPTION:
The study consists of 2 parts, Part A and Part B. Part A consists of the dose escalation cohorts and will include patients with metastatic castration resistant prostate cancer (mCRPC) or metastatic castration-sensitive prostate cancer (mCSPC); Part B consists of dose expansion cohorts and will include patients with mCSPC only.

Part A comprises 4 individual arms each evaluating the safety, tolerability, and preliminary efficacy of AZD5305 in combination with a specific new hormonal agent (NHA). Part B comprises up to 4 individual arms (arms to be opened at Sponsor's discretion) each investigating the preliminary efficacy and aims to further build on the safety data for the combination of AZD5305 with a specific NHA.

Approximately 783 patients will be enrolled and screened to ensure the required number of evaluable patients in each part and arm are enrolled. For Part A, 356 patients may be screened to obtain up to approximately 308 patients that can be assigned to study treatments across all study arms (1 to 4). For Part B dose expansion cohorts, up to 427 patients may be screened to obtain up to approximately 360 patients that can be assigned to study treatments across all study arms (1 to 4).

Study treatment administration will continue until disease progression, initiation of alternative anticancer therapy, unacceptable toxicity, withdrawal of consent, or other reasons to discontinue study treatment occur.

ELIGIBILITY:
Inclusion Criteria:

For whole study:

* Age ≥ 18 at the time of screening.
* Histologically confirmed diagnosis of metastatic prostate cancer.
* Candidate for treatment with enzalutamide, abiraterone acetate, darolutamide or apalutamide with documented current evidence of metastatic prostate cancer.
* Surgically or medically castrated.
* Adequate organ and marrow function.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS): 0-1 with no deterioration over the previous 2 weeks.
* Life expectancy ≥ 16 weeks.
* Non-sterilized male patients who are sexually active with a female partner of childbearing potential must use a condom with spermicide from screening to approximately 6 months after the last dose of study treatment .

For Patients Recruited Specifically to tumour Pharmacodynamic Cohorts:

• Patients must have at least 1 tumour suitable for paired biopsies

For Part A:

• Patients with Metastatic Castrate ion-Resistant Prostate Cancer (mCRPC) or Metastatic Castration Sensitive Prostate Cancer (mCSPC).

For Part B:

• Patients must have mCSPC (de novo or recurrent) with a baseline PSA value of ≥ 0.2 ng/mL

Exclusion Criteria:

For Part A mCRPC patients only:

* Any previous treatment with a new hormonal agent (NHA), poly (adenosine diphosphateribose) polymerase inhibitor (PARPi), Lutetium prostate-specific membrane antigen (Lu-PSMA), platinum chemotherapy
* Patients recruited to the PDc cohorts should not have received a prior use of new hormonal agents (NHA).

For Part A and Part B mCSPC Patients:

* Any previous treatment with a PARPi, platinum, NHA, Immuno-oncology (IO), radiopharmaceutical therapy, or prior treatment with docetaxel in mCSPC setting.
* Concomitant use of medications or herbal supplements known to be:

  1. Strong and moderate CYP3A4 inducers/inhibitors (applies for all arms)
  2. For Arm 1 (enzalutamide) patients: Strong CYP2C8 inhibitors
  3. For Arm 3 (darolutamide) patients: Strong P-glycoprotein inducers
* Concomitant use of drugs that are known to prolong or shorten QT and have a known risk of Torsades de Pointes.
* Treatment with any of the following:

  1. Any investigational agents or study interventions from a previous clinical study within 5 half lives or 3 weeks (whichever is longer) of the first dose of study treatment.
  2. Any other anticancer treatment within the following time periods prior to the first dose of study treatment: (i) Cytotoxic and non-cytotoxic treatment: 3 weeks or 5 half-lives (whichever is shorter). (ii) Biological products including immuno-oncology agents: 4 weeks before enrolment.
  3. Any live virus or bacterial vaccine within 28 days of the first dose of study treatment.
* Any concurrent anticancer therapy or concurrent use of prohibited medications.
* Major surgery within 4 weeks prior to the first dose of study treatment.
* Radiotherapy with a wide field of radiation within 4 weeks or radiotherapy with a limited field of radiation for palliation within 2 weeks of the first dose of study treatment.
* With the exception of alopecia, and peripheral neuropathy; any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 at the time of study enrolment.
* Any history of persisting (> 2 weeks) severe pancytopenia.
* Spinal cord compression, or brain metastases unless asymptomatic and treated and stable.
* Any evidence of severe or uncontrolled systemic diseases, including, active bleeding diatheses, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV).
* Patients with any known predisposition to bleeding (eg, active peptic ulceration, recent [within 6 months] haemorrhagic stroke, proliferative diabetic retinopathy.
* Any clinically significant cardiac disorders including QT prolongation, abnormal electrocardiogram (ECG).
* Any clinically significant cardiovascular diseases including symptomatic heart failure, uncontrolled hypertension, acute coronary syndrome, cardiomyopathy, valvular heart disease, atrial fibrillation, stroke.
* Patients with history of myelodysplastic syndrome (MDS)/ acute myeloid leukaemia (AML).
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection.
* Known allergy or hypersensitivity to investigational product(s) or any of the excipients of the investigational product(s).
* Any condition that would interfere with evaluation of the study treatment or interpretation of patient safety or study results.
* Uncontrolled intercurrent illness within the last 12 months, including but not limited to, active interstitial lung disease, serious chronic gastrointestinal (GI) conditions associated with diarrhoea, or psychiatric illness/social situations
* History of another primary malignancy except for malignancy treated with curative intent with no known active disease within 3 years before the first dose of study treatment and of low potential risk for recurrence.
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
* Arm 1 (Enzalutamide) and Arm 4 (Apalutamide): History of seizure or any condition that may predispose to seizure (eg, prior cortical stroke, significant brain trauma).
* Arm 2 (Abiraterone acetate) only: (i) Active infection or other medical condition that would contraindicate the use of systemic steroids (prednisone/prednisolone). (ii) Low serum potassium (< 3.5 mmol/L). (iii) History of uncontrolled pituitary or adrenal dysfunction.
* Arm 4 (Apalutamide): (i) Moderate or severe skin conditions or diseases that could affect the skin (eg. scleroderma, lupus). (ii) Any skin or medical condition that in the Investigator's opinion could increase the risk of skin toxicity.

Ages: 18 Years to 130 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2031-04-11 (Estimated); Study Completion 2031-04-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Adverse Events and Serious Adverse Events | Up to post treatment follow-up (28 days after last dose) [assessed up to 2.3 years]
  Number of patients with adverse events and with serious adverse events including abnormal clinical observations, abnormal ECG parameters, abnormal laboratory assessments and abnormal vital signs that changed from baseline will be assessed.
Part A: Number of patients with Dose Limiting Toxicities (DLTs) | For Arm 1: 35 days, For Arm 2 and 3: 28 days
  To assess the safety and tolerability of AZD5305 when given in combination with NHA.

SECONDARY OUTCOMES:
Area Under the concentration Curve (AUC) of AZD5305 | At the end of Cycle 0 (Cycle 0 is of 7 days)
  To characterise the PK (AUC) of AZD5305 at steady state after multiple dosing of AZD5305 monotherapy.
Maximum plasma concentration (Cmax) of AZD5305 | At the end of Cycle 0 (Cycle 0 is of 7 days)
  To characterise the PK (Cmax) of AZD5305 at steady state after multiple dosing of AZD5305 monotherapy.
Time to maximum concentration (tmax) of AZD5305 | At the end of Cycle 0 (Cycle 0 is of 7 days)
  To characterise the PK (tmax) of AZD5305 at steady state after multiple dosing of AZD5305 monotherapy.
AUC of AZD5305 | Arm 1: At Cycle 1 Day 1, Cycle 1 Day 22, Cycle 2 Day 1, Cycle 2 Day 2, Cycle 2 Day 8, and Cycle 3 Day 1; Arm 2 and 3: At Cycle 1 Day 1, Cycle 1 Day 15 and Cycle 2 Day 1 (Each Cycle is of 28 days)
  To characterise the PK (AUC) of AZD5305 following oral dose administration of AZD5305 in combination with NHA.
Cmax of AZD5305 | Arm 1: At Cycle 1 Day 1, Cycle 1 Day 22, Cycle 2 Day 1, Cycle 2 Day 2, Cycle 2 Day 8, and Cycle 3 Day 1; Arm 2 and 3: At Cycle 1 Day 1, Cycle 1 Day 15 and Cycle 2 Day 1 (Each Cycle is of 28 days)
  To characterise the PK (Cmax) of AZD5305 following oral dose administration of AZD5305 in combination with NHA.
tmax of AZD5305 | Arm 1: At Cycle 1 Day 1, Cycle 1 Day 22, Cycle 2 Day 1, Cycle 2 Day 2, Cycle 2 Day 8, and Cycle 3 Day 1; Arm 2 and 3: At Cycle 1 Day 1, Cycle 1 Day 15 and Cycle 2 Day 1 (Each Cycle is of 28 days)
  To characterise the PK (tmax) of AZD5305 following oral dose administration of AZD5305 in combination with NHA.
Objective response rate (ORR) | From Screening (Day -28) to confirmed disease progression [assessed up to 2.3 years]
  To assess the preliminary antitumour activity of AZD5305 in combination with NHA. ORR will be assessed as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 (soft tissue) and Prostate Cancer Clinical Trials Working Group 3 (PCWG3) and is defined as the percentage of patients who have a confirmed visit response of complete response (CR) or partial response (PR) in their soft tissue disease and no disease progression in their bone scan.
Duration of response (DoR) | From Screening (Day -28) to confirmed disease progression [assessed up to 2.3 years]
  To assess the preliminary antitumour activity of AZD5305 in combination with NHA. DoR is defined as the time from the date of first documented response (which is subsequently confirmed) until date of documented progression or death in the absence of progressive disease (PD).
Time to response (TTR) | From Screening (Day -28) to confirmed disease progression [assessed up to 2.3 years]
  To assess the preliminary antitumour activity of AZD5305 in combination with NHA. TTR is defined as the time from first dose until the first documentation of a subsequently confirmed objective response.
Radiographic progression-free survival (rPFS) | From Screening (Day -28), 12 months, 24 months and up to confirmed disease progression [assessed up to 2.3 years]
  To assess the preliminary antitumour activity of AZD5305 in combination with NHA. rPFS is defined as the time from start of first treatment until progression as per RECIST v1.1 (soft tissue) and PCWG3 criteria (bone) or death from any cause.
Percentage change in tumour size | From Screening (Day -28) to confirmed disease progression [assessed up to 2.3 years]
  To assess the preliminary antitumour activity of AZD5305 in combination with NHA. Percentage change in tumour size will be determined for patients with measurable disease at baseline.
Number of patients with ≥ 50% prostate-specific antigen (PSA) decrease from baseline | From Screening (Day -28) to confirmed disease progression [assessed up to 2.3 years]
  To assess the preliminary antitumour activity of AZD5305 in combination with NHA.
Number of patients with ≥ 90% prostate-specific antigen (PSA) decrease from baseline | From Screening (Day -28) to confirmed disease progression [assessed up to 2.3 years]
  To assess the preliminary antitumour activity of AZD5305 in combination with NHA.
Part B: Number of patients with undetectable PSA (< 0.2 ng/mL) | 3, 6, 9 and 12 months
  To assess the preliminary antitumour activity of AZD5305 in combination with NHA.
PSA Progression-free survival | 6, 12, 18, 24 and 30 months
  To assess the preliminary antitumour activity of AZD5305 in combination with NHA.
AUC of Enzalutamide | At Cycle 1 Day 22, Cycle 2 Day 1, Cycle 2 Day 2, Cycle 2 Day 8 and Cycle 3 Day 1 (Each Cycle is of 28 days)
  To characterize the PK (AUC) of Enzalutamide in plasma at steady state when given orally in combination with AZD5305
Cmax of Enzalutamide | At Cycle 1 Day 22, Cycle 2 Day 1, Cycle 2 Day 2, Cycle 2 Day 8 and Cycle 3 Day 1 (Each Cycle is of 28 days)
  To characterize the PK (Cmax) of Enzalutamide in plasma at steady state when given orally in combination with AZD5305
tmax of Enzalutamide | At Cycle 1 Day 22, Cycle 2 Day 1, Cycle 2 Day 2, Cycle 2 Day 8 and Cycle 3 Day 1 (Each Cycle is of 28 days)
  To characterize the PK (tmax) of Enzalutamide in plasma at steady state when given orally in combination with AZD5305
AUC of Apalutamide | At Cycle 1 Day 22, Cycle 2 Day 1, Cycle 2 Day 2, Cycle 2 Day 8 and Cycle 3 Day 1 (Each Cycle is of 28 days)
  To characterize the PK (AUC) of Apalutamide in plasma at steady state when given orally in combination with AZD5305
Cmax of Apalutamide | At Cycle 1 Day 22, Cycle 2 Day 1, Cycle 2 Day 2, Cycle 2 Day 8 and Cycle 3 Day 1 (Each Cycle is of 28 days)
  To characterize the PK (Cmax) of Apalutamide in plasma at steady state when given orally in combination with AZD5305
tmax of Apalutamide | At Cycle 1 Day 22, Cycle 2 Day 1, Cycle 2 Day 2, Cycle 2 Day 8 and Cycle 3 Day 1 (Each Cycle is of 28 days)
  To characterize the PK (tmax) of Apalutamide in plasma at steady state when given orally in combination with AZD5305
Part B: Homologous recombination repair gene mutation (HRRRm) | From Screening (Day -28) to confirmed disease progression [assessed up to 2.3 years]
  To investigate HRRm (including BRCA1/2) and their relationship with clinical response

CONTACTS AND LOCATIONS:
Locations (18):
- United States (4):
  - Research Site, Detroit, Michigan
  - Research Site, Syracuse, New York
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Houston, Texas
- Australia (6):
  - Research Site, Camperdown
  - Research Site, Darlinghurst
  - Research Site, East Melbourne
  - Research Site, Heidelberg
  - Research Site, Melbourne
  - Research Site, St Leonards
- Italy (4):
  - Research Site, Candiolo
  - Research Site, Milan
  - Research Site, Orbassano
  - Research Site, Padua
- United Kingdom (4):
  - Research Site, Cambridge
  - Research Site, Glasgow
  - Research Site, Manchester
  - Research Site, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home